CLINICAL TRIAL: NCT01510171
Title: Rapid Activity of Platelet Inhibitor Drugs Study
Acronym: RAPID
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Careggi Hospital (Other)
Responsible Party: Principal Investigator, David Antoniucci, Head Division of Invasive Cardiology, Careggi Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RAPID
Record Dates: First submitted 2012-01-11; First posted 2012-01-13 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2014-09

CONDITIONS: ST-segment Elevation Myocardial Infarction
Keywords: platelet inhibitor; ST-segment elevation myocardial infarction; stent; prasugrel; ticagrelor
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — Prasugrel Hydrochloride; Ticagrelor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Prasugrel loading dose (Active Comparator)
  Interventions: Drug: Prasugrel
- Ticagrelor Loading dose (Active Comparator)
  Interventions: Drug: Ticagrelor

INTERVENTIONS:
Drug: Prasugrel — 25 patients with STEMI undergoing PPCI with bivalirudin (GP IIb/IIIa not allowed ) will be enrolled to receive 60 mg Prasugrel loading dose before PPCI. The loading dose will be performed as soon as possible in the Emergency Room or in the Cath Lab. In the case of vomit in the 2 hours after drug loading dose a new loading dose will be administered.
  Arms: Prasugrel loading dose
Drug: Ticagrelor — 25 patients with STEMI undergoing PPCI with bivalirudin (GP IIb/IIIa not allowed ) will be enrolled to receive 180 Ticagrelor loading dose before PPCI. The loading dose will be performed as soon as possible in the Emergency Room or in the Cath Lab. In the case of vomit in the 2 hours after drug loading dose a new loading dose will be administered.
  Arms: Ticagrelor Loading dose

SUMMARY:
The aim of the RAPID study is to assess the rapid onset of action of the 2 novel oral antiplatelet agents, Prasugrel and Ticagrelor, in 50 patients with STEMI undergoing PPCI with bivalirudin monotherapy.

DETAILED DESCRIPTION:
Fifty consecutive patients with STEMI undergoing PPCI with bivalirudin (GP IIb/IIIa not allowed ) will be randomized to receive 60 mg Prasugrel loading dose (n= 25) or 180 Ticagrelor loading dose (n= 25) before PPCI. The loading dose will be performed as soon as possible in the Emergency Room or in the Cath Lab. In the case of vomit in the 2 hours after drug loading dose a new loading dose will be administered. All interventions will be performed by the femoral approach according to current standards. The use of thrombectomy before infarct-related artery stenting, of everolimus eluting stent and of closure devices will be strongly encouraged. Bivalirudin will be administered as a bolus 0.75 mg/kg followed by 1.75 mg/kg/h infusion during PCI. After PCI a reduced bivalirudin infusion of 0.25 mg/kg/h for 4 hours will be allowed. Dual antiplatelet therapy (100 mg aspirin associated with 5 or 10 mg Prasugrel or 180 mg Ticagrelor) will be recommended for 12 months.

Residual platelet reactivity will be assessed in all patients at baseline (time of loading dose), and after 2, 4, 8 and 12 hours by a point-of-care test VerifyNow bedside available in the Intensive cardiac care Unit. High residual platelet reactivity will be defined as a Platelet Reactivity Units (PRU) > 240 by VerifyNow. At the same time point, Activated Clotting Time (ACT) will be also assessed. Follow-up will be performed by outpatient visits or telephone interviews at 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Patients presenting within 12 hours from the onset of symptoms with STEMI
2. Informed, written consent

Exclusion Criteria:

1. Age < 18 years
2. Active bleeding; bleeding diathesis; coagulopathy
3. History of gastrointestinal or genitourinary bleeding <2 months
4. Major surgery in the last 6 weeks
5. History of intracranial bleeding or structural abnormalities
6. Suspected aortic dissection
7. Any previous TIA/stroke
8. Administration in the week before the index event of clopidogrel, ticlopidine, prasugrel, ticagrelor, thrombolytics, bivalirudin, low-molecular weight heparin or fondaparinux, GPI.
9. Known relevant hematological deviations: Hb <10 g/dl, Platelet count <100x10^9/l
10. Use of coumadin derivatives within the last 7 days
11. Chronic therapy with prasugrel or ticagrelor
12. Known malignancies or other comorbid conditions with life expectancy <1 year
13. Known severe liver disease, severe renal failure
14. Known allergy to the study medications
15. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-01; Primary Completion 2012-06 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Residual platelet reactivity by VerifyNow | 2 hours
  Residual platelet reactivity will be assessed in all patients at baseline (time of loading dose), and after 2 hours by a point-of-care test VerifyNow bedside available in the Intensive cardiac care Unit.

SECONDARY OUTCOMES:
High residual platelet reactivity | 2,4,8,12 hours
  High residual platelet reactivity will be defined as a Platelet Reactivity Units (PRU) > 240 by VerifyNow.

CONTACTS AND LOCATIONS:
Overall Officials: David Antoniucci, MD, Principal Investigator — Careggi Hospital, Division of Invasive Cardiology
Locations (1):
- Careggi Hospital, Florence, Italy

REFERENCES:
- [Derived] Parodi G, Valenti R, Bellandi B, Migliorini A, Marcucci R, Comito V, Carrabba N, Santini A, Gensini GF, Abbate R, Antoniucci D. Comparison of prasugrel and ticagrelor loading doses in ST-segment elevation myocardial infarction patients: RAPID (Rapid Activity of Platelet Inhibitor Drugs) primary PCI study. J Am Coll Cardiol. 2013 Apr 16;61(15):1601-6. doi: 10.1016/j.jacc.2013.01.024. Epub 2013 Mar 22. PMID 23500251